CLINICAL TRIAL: NCT05976243
Title: A 52-week Multi-center, Randomized, Double-blind, Placebo Controlled, Basket Study With an Open-label Extension to Investigate the Efficacy, Safety, and Tolerability of Remibrutinib (LOU064) in Chronic Inducible Urticaria (CINDU) in Adults Inadequately Controlled by H1-antihistamines
Brief Title: A Study to Investigate Efficacy, Safety, and Tolerability of Remibrutinib Compared With Placebo in Adults With CINDU Inadequately Controlled by H1-antihistamines
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLOU064M12301; 2023-505739-12-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Inducible Urticaria
Keywords: CINDU; Chronic inducible urticaria; BTK; remibrutinib; symptomatic dermographsim; cold urticaria; cholinergic urticaria
MeSH Terms: conditions — Chronic Inducible Urticaria; Cold Urticaria | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This masking applies to the core period. There is no masking in the open-label extension (OLE).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Remibrutinib, symptomatic dermographism group (Experimental): Remibrutinib oral twice daily in participants with symptomatic dermographism
  Interventions: Drug: Remibrutinib
- Placebo, symptomatic dermographism group (Placebo Comparator): Placebo oral twice daily, symptomatic dermographism
  Interventions: Other: Placebo
- Remibrutinib, cold urticaria group (Experimental): Remibrutinib oral twice daily, cold urticaria
  Interventions: Drug: Remibrutinib
- Placebo, cold urticaria group (Placebo Comparator): Placebo oral twice daily, cold urticaria
  Interventions: Other: Placebo
- Remibrutinib, cholinergic urticaria group (Experimental): Remibrutinib oral twice daily, cholinergic urticaria
  Interventions: Drug: Remibrutinib
- Placebo, cholinergic urticaria (Placebo Comparator): Placebo oral twice daily, cholinergic urticaria
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Remibrutinib — Remibrutinib treated groups and arms
  Arms: Remibrutinib, cholinergic urticaria group; Remibrutinib, cold urticaria group; Remibrutinib, symptomatic dermographism group
Other: Placebo — Placebo treated groups and arms
  Arms: Placebo, cholinergic urticaria; Placebo, cold urticaria group; Placebo, symptomatic dermographism group

SUMMARY:
This is a Phase 3, parallel group, placebo-controlled, double-blind, confirmatory study in patients with CINDU, with an optional Open-label Extension (OLE).

The purpose of the core period (52 weeks of treatment) of this study is to evaluate the efficacy, safety, and tolerability of remibrutinib (LOU064) vs. placebo in adults suffering from CINDU inadequately controlled by H1-antihistamines (H1-AHs).

The purpose of the OLE period is to collect long-term efficacy, safety, and tolerability data on remibrutinib in participants after having completed the Core period

DETAILED DESCRIPTION:
This study consists of a core and extension periods.

The Core period (6 arms) has a total duration of up to 60 weeks including a double-blind placebo-controlled treatment period until Week 24 followed by open-label treatment with remibrutinib up to Week 52. The primary endpoint for all CINDU subtypes is assessed at Week 12.

The Core period consists of:

* Screening period (up to 4 weeks): During the screening period, participants who have provided informed consent will be assessed for study eligibility.
* Double-blind, placebo-controlled treatment period (24 weeks): 24 weeks of double-blind treatment with remibrutinib or placebo.
* Open-label treatment period (28 weeks): 28 weeks of open-label treatment with remibrutinib.
* Follow-up period: 4 weeks of treatment free follow-up. The open-label extension period consists of observation and treatment period. At the end of the core period of the study, if participants continue to experience symptoms, they will transition to the treatment period in OLE. If they do not experience symtpoms they will transition to the observation period in the OLE.

The duration of the Open-label Extension period will be approximately 3 years where participants can switch from observation to treatment depending on if they start developing symptoms. Only those participants participating in the Open-label Extension Treatment period will receive remibrutinib. The participants in the Open-label Extension Observation period will not receive remibrutinib

ELIGIBILITY:
Inclusion Criteria for core period:

1. Male and female participants ≥18 years of age at the time of signing of the ICFs
2. Confirmed CINDU diagnosis (as per guidelines) for symptomatic dermographism, cold urticaria or cholinergic urticaria for ≥ 4 months (defined as onset of CINDU with supporting documentation (e.g medical record, clinical history, photographs)) and inadequate control with H1-AH at local label approved doses at the time of randomization
3. The following response to the provocation test for each subtype is required at the randomization visit :

   * Symptomatic Dermographism: A Total Fric Score of ≥3 using the FricTest® 4.0 and a numerical rating scale score of ≥5 for itch after the provocation test.
   * Cold Urticaria: A Critical Threshold Temperature of ≥15°C using the TempTest® 4.0 and a numerical rating scale score of ≥5 for itch after the provocation test.
   * Cholinergic Urticaria: A physician global assessment of severity of hives ≥ 2 using the Pulse-controlled ergometry test and a numerical rating scale score of ≥5 for itch after the provocation test.
4. Cold Urticaria: Positive ice-cube test resulting in hives at the provocation site for participants at Screening.
5. Cholinergic urticaria: Participants must show sweating in performing the pulse-controlled ergometry test on day of randomization. Participants with anhidrosis must not be included.

Inclusion criteria for the OLE:

1. Participants who have completed the Core period up to Week 52 and are willing to enter the OLE period

   Exclusion Criteria for core period:
   * 1. Previous use of remibrutinib or other BTK inhibitors.
2. Participants who have concomitant CSU at screening. Participants with resolved CSU at the time of screening can be included in the study.
3. Participants who have a familial form (e.g familial cold autoinflammatory syndrome, familial cold urticaria) of the target CINDU that is being considered for the participant's inclusion in this study.
4. Participants having a more defined other form of inducible urticaria than the target CINDU that is being considered for the participant's inclusion in this study.
5. Diseases, other than chronic inducible urticaria, with urticaria or angioedema symptoms including but not limited to urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema
6. Any other skin disease associated with chronic itching that might influence, in the investigator's opinion, the study evaluations and results (e.g., atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, etc.) or skin diseases associated with only wheals and no itch e.g asymptomatic dermographism

There are no exclusion criteria for OLE

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with complete response in Total Fric Score; symptomatic dermographism | Week 12
  Total Fric score (a scale from 0-4 where a positive response with all of the four pins is TFS = 4, while a positive response with only one pin - the largest pin is TFS = 1)
Proportion of participants with complete response in critical temperature threshold; cold urticaria | Week 12
  The Temptest is used to induce itch and hives in participants with cold urticaria. Critical temperature threshold (CTT), as measured by the Temptest, determines the highest temperature that induces symptoms.
Proportion of participants with itch numerical rating scale =0; cholinergic urticaria | Week 12
  Itch numerical rating scale, a scale from 0 to 10
  Patients are asked to rate itching severity based on the worst level of itching in the past 24 h using an 11-point scale from 0 ("no itch") to 10 ("worst itch imaginable")

SECONDARY OUTCOMES:
Change from baseline in Total Fric score; symptomatic dermographism | Week 12
  Total Fric score, a scale from 0-4 where a positive response with all four pins is TFS=4, while a positive only 1 pin - the largest pin is TFS=1
Change from baseline in criticial temperature threshold following Temptest; cold urticaria | Week 12
  Critical temperature threshold, as measured by the Temptest, determines the highest temperature that induces symptoms
Change from baseline in itch numerical rating scale; cholinergic urticaria | Week 12
  Itch numerical rating scale (NRS), scale from 0 to 10. 0 ("no itch") to 10 ("worst imaginable itch").
proportion of participants with Physician Global Assessment (PGA) severity of hives =0; cholinergic urticaria | Week 12
  Physician global assessment of severity of hives. This assessment is scored 0 to 4 with 0=no hives, 1=mild hives, 2=moderate hives, 3=severe hives and 4=very severe hives
Proportion of participants with complete response in TFS; symptomatic dermographism | Week 24
  Total Fric score (a scale from 0-4 where a positive response with all of the four pins is TFS = 4, while a positive response with only one pin - the largest pin is TFS = 1)
Proportion of participants with complete response in Critical Temperature threshold; cold urticaria | Week 24
  Critical Temperature Threshold, as measured by the Temptest, is the highest temperature that induces symptoms
Proportion of participants with complete response in itch numerical rating scale; cholinergic urticaria | Week 24
  Itch numerical rating scale (NRS), scale from 0 to 10. 0 ("no itch") to 10 ("worst imaginable itch").
Change from baseline in itch numerical rating scale in participants with symptomatic dermographism | Week 12
  Itch numerical rating scale (NRS), scale from 0 to 10. 0 ("no itch") to 10 ("worst imaginable itch").
Change from baseline in itch numerical rating scale in participants with cold urticaria | Week 12
  Itch numerical rating scale (NRS), scale from 0 to 10. 0 ("no itch") to 10 ("worst imaginable itch").
Proportion of participants with complete response in Total Fric score; symptomatic dermographism | Week 2
  Total Fric score (a scale from 0-4 where a positive response with all of the four pins is TFS = 4, while a positive response with only one pin - the largest pin is TFS = 1)
Proportion of participants with complete response in Critical Temperature Threshold; cold urticaria | Week 2
  Critical temperature threshold (CTT), as measured by the Temptest, determines the highest temperature that induces symptoms.
Proportion of participants with itch NRS=0; cholinergic urticaria | Week 2
  Itch numerical rating scale (NRS), scale from 0 to 10. 0 ("no itch") to 10 ("worst imaginable itch").
Change from baseline in TFS in participants with symptomatic dermographism | Week 2
  Total Fric score (a scale from 0-4 where a positive response with all of the four pins is TFS = 4, while a positive response with only one pin - the largest pin is TFS = 1)
Change from baseline in Critical Temperature Threshold in participants with cold urticaria | Week 2
  Critical temperature threshold (CTT), as measured by the Temptest, determines the highest temperature that induces symptoms.
Change from baseline in itch NRS in participants with cholinergic urticaria | Week 2
  Itch numerical rating scale (NRS), scale from 0 to 10. 0 ("no itch") to 10 ("worst imaginable itch").
Change from baseline in itch NRS in participants with symptomatic dermographism | Week 2
  Total Fric score (a scale from 0-4 where a positive response with all of the four pins is TFS = 4, while a positive response with only one pin - the largest pin is TFS = 1)
Change from baseline in itch NRS in participants with cold urticaria | Week 2
  Itch numerical rating scale (NRS), scale from 0 to 10. 0 ("no itch") to 10 ("worst imaginable itch").
Proportion of participants with cholinergic urticaria with PGA=0 | Week 2
  Physician global assessment of severity of hives is a 4-point scale (0 = no active disease, 1 = mild disease, 2 = moderate disease, 3 = severe disease).
Change from baseline in weekly most bothersome symptom NRS score on the USDD | Week 12
  Urtricara symptom daily diary (USDD). This daily diary records if the participant experiences any symptoms or avoided the triggers
Proportion of participants with DLQI=0-1 | Week 12
  The Dermatology Life Quality Index (DLQI) is a 10-item dermatology-specific quality of life (QoL) measure. Subjects rate their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives thinking about the previous 7 days. An overall score is calculated and ranges from 0 to 30 (higher score meaning worse disease-related QoL). A DLQI score of 0 or 1 means that there is no impact of a skin disease on the patient's life.
Occurrence of treatment emergent adverse events and serious adverse events during the study | Week 52
  Treatment emergent adverse events and serious adverse events are those that occur at any time only after treatment has started

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (128):
- United States (25):
  - Allervie Clinical Research, Birmingham, Alabama
  - Acuro Research Inc, Little Rock, Arkansas
  - Kern Research, Bakersfield, California
  - Allergy and Asthma Specialists Group, Huntington Beach, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Asthma and Allergy Associates P C, Colorado Springs, Colorado
  - Florida Ctr Allergy Asthma Research, Aventura, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Univ of South Florida Asthma Allergy and Immunology CRU, Tampa, Florida
  - Aeroallergy Research Laboratories, Savannah, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Endeavor Health, Glenview, Illinois
  - Asthma and Allergy Center of Chicago S C, River Forest, Illinois
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Allergy and Asthma Specialist P S C, Owensboro, Kentucky
  - John Hopkins University, Baltimore, Maryland
  - Allergy Asthma and Clinical Research, Oklahoma City, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research LLS, North Charleston, South Carolina
  - PanAmerican Clinical Research, Brownsville, Texas
  - Western Sky Medical Research, El Paso, Texas
  - RFSA Dermatology, San Antonio, Texas
  - STAAMP Research LLC, San Antonio, Texas
  - Complete Dermatology, Sugar Land, Texas
  - Allergy Associates of Utah, Sandy City, Utah
- Argentina (4):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, CABA
- Australia (3):
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Carlton, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
- Brazil (3):
  - Novartis Investigative Site, Alphaville Barueri, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, Sorocaba, São Paulo
- Canada (3):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Trois-Rivières, Quebec
- China (14):
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Yiwu, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Barranquilla, Atlántico, Colombia
- France (8):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
- Germany (7):
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (3):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Debrecen, Hajdú-Bihar
  - Novartis Investigative Site, Szolnok, Jász-Nagykun-Szolnok
- India (3):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (3):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Japan (13):
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Ohtsu, Shiga
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Shimotsuga Gun, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Hiroshima
- Malaysia (3):
  - Novartis Investigative Site, Muar town, Johor
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, George Town, Pulau Pinang
- Novartis Investigative Site, Utrecht, Netherlands
- Poland (2):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Warsaw
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Vila Nova de Gaia
- Novartis Investigative Site, Bucharest, District 2, Romania
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (3):
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Trnava
  - Novartis Investigative Site, Žilina
- South Korea (2):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Santiago, A Coruna
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Sakarya, Adapazari
  - Novartis Investigative Site, Istanbul, Basaksehir
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Istanbul, Uskudar
- Novartis Investigative Site, Oxford, United Kingdom
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com